CLINICAL TRIAL: NCT00588211
Title: Measurement of Cancer-Related Risk Perception in Smokers
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Adelphi University (Other); Queen's Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 01-121; CA93182
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Cancer Related-Risks; Risk Perception; Survey; Focus Group
Keywords: Cancer related-Risks; Risk Perception; Survey; Focus Group; Smoking cessation; tobacco
MeSH Terms: conditions — Smoking Cessation | interventions — Interviews as Topic; Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (4):
- 1: We will recruit fifteen New York University College of Dentistry (NYUCD) clinic patients who report current tobacco use.
  Interventions: Behavioral: Interviews
- 2: Second, we will recruit thirty dental clinic smokers (10 per day for 3 days) from the NYUCD waiting room.
  Interventions: Behavioral: focus group
- 3: Third, we will survey 200 student participants from Adelphi University.
  Interventions: Behavioral: Survey
- 4: Queens Hospital Center with 800 patients.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Interviews — 45-minute individual interviews after the conclusion of their dental appointment
  Groups: 1
Behavioral: focus group — A focus group of the preliminary cancer-related risk perception item pool.
  Groups: 2
Behavioral: Survey — Quantitative item analysis of the final item pool.
  Groups: 3
Behavioral: Survey — A second confirmatory factor analysis.
  Groups: 4

SUMMARY:
The purpose of this study is to develop an accurate way of measuring people's thoughts about cancer risk. The researchers at the Queens Hospital Center, Memorial Sloan-Kettering Cancer Center and Adelphi University are working together to design a new measure. Findings from this study will help us find new ways to help people avoid cancer.

DETAILED DESCRIPTION:
The goal of the study is to develop and provide initial evidence for the reliability and validity of a measure of cancer-related risk perception. As such, the primary outcomes of the study will be initial construct validity (convergent validity and discriminant validity) of the proposed scale as evidenced by correlations of this test with other tests that vary in the degree of association to the proposed construct of cancer-related risk perception. It is anticipated that the cancer-related risk perception scale will correlate most highly (.50-.60) with measures of tobacco and environmental risk exposures, readiness to quit smoking, and family cancer history.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be >= to 18 years of age
* For recruitment at Adelphi University: Speak English
* For recruitment at Queens Hospital Center: Speak English
* For recruitment at Queens Hospital Center: Must be a Queens Hospital Center Patient

Exclusion Criteria:

* Patients who have a history of colorectal cancer at the Queens Hospital Center
* Patients who cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * clinic patients Queens Hospital Center
  * students participants from Adelphi University
Sampling Method: Non-Probability Sample
Enrollment: 1514 (Actual)
Dates: Start 2001-09; Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Develop a comprehensive "blueprint," or description of the cancer-related risk perception construct; to use it to generate a cancer-related risk perception item pool; conduct an analysis of the generated items | 3 years

SECONDARY OUTCOMES:
to establish initial evidence for scale reliability and validity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Hay, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Queens Hospital Center, Jamaica, New York
  - New York University, College of Dentistry, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Adelphi University, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org